CLINICAL TRIAL: NCT06823726
Title: Efficacy and Safety of a 12-Week Taekwondo Training Program in Patients With Ankylosing Spondylitis and Axial Spondyloarthritis: A Randomized Controlled Trial
Brief Title: Taekwondo for Axial Spondyloarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Nam, Seoung Wan, Assistant Professor, Division of Rheumatology, Department of Internal Medicine, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR324115
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis
Keywords: Taekwondo; Ankylosing Spondylitis; Axial Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-blind, parallel-group, exploratory pilot randomized controlled trial to evaluate the efficacy and safety of a 12-week Taekwondo training program in patients with ankylosing spondylitis and axial spondyloarthritis.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taekwondo training group (Experimental): Participants will undergo a 12-week Taekwondo training program, consisting of three 60-minute sessions per week.
  Interventions: Other: 12-week Taekwondo training
- Control group (No Intervention): Participants will maintain their usual daily activities for 12 weeks without any structured exercise intervention.

INTERVENTIONS:
Other: 12-week Taekwondo training — 12-week structured Taekwondo training program under the supervision of qualified instructors following a standardized protocol.
  Frequency: 3 sessions per week Session Length: 60 minutes per session
  Arms: Taekwondo training group

SUMMARY:
The goal of this clinical trial is to learn if Taekwondo training works to help adults with ankylosing spondylitis and axial spondyloarthritis. It will also learn about the safety of Taekwondo training for these adults.

The main questions are as follows:

* Will Taekwondo training affect disease activity, functional improvement, and quality of life?
* Will there be a difference between adults who participate in Taekwondo training and adults who continue with their usual treatment?
* Is Taekwondo training safe for adults with ankylosing spondylitis and axial spondyloarthritis, and will it be an appropriate exercise for these adults?
* Is there a possibility to develop a structured Taekwondo-based exercise program for adults with musculoskeletal disorders?

Participants will:

* Be a part of the Taekwondo training group or the control group for 12 weeks (where the control group will later participate in the same 12 week Taekwondo for comparison)
* Be assessed within 2 weeks before the start of the training
* Be assessed within 1 week after completing the training

DETAILED DESCRIPTION:
This study is designed as a single-blind, parallel-group, exploratory pilot randomized controlled trial to evaluate the efficacy and safety of a 12-week Taekwondo training program in patients with ankylosing spondylitis and axial spondyloarthritis.

1) Total Taekwondo Intervention Period: 24 Weeks

1. Initial 12 weeks: Comparison between the Taekwondo training group and the control group in an RCT.
2. Post-RCT 12 weeks: The control group receives the same Taekwondo training, allowing for a pre- and post-intervention comparison.

2) Assessment Time Points

1. Baseline (Pre-Intervention): Within 2 weeks before the start of the 12-week Taekwondo training.
2. End of RCT (Post-Intervention): Within 1 week after completing the initial 12-week Taekwondo training.

   The primary effects of the intervention will be assessed through comparisons between the Taekwondo training group and the control group.
3. End of Control Group Intervention: Within 1 week after completing the 12-week Taekwondo training in the control group.

Pre- and post-intervention comparisons will be conducted for the control group. 3) Group Composition

1. Taekwondo Training Group: Participates in a structured 12-week Taekwondo training program during the RCT period.
2. Control Group: Maintains usual daily activities for the initial 12 weeks, followed by participation in the same 12-week Taekwondo training program.

4) Blinding Procedure

1. Evaluator Blinding: The assessors conducting the outcome evaluations will remain blinded to the intervention status of participants to ensure unbiased assessments. All evaluations will be performed in a neutral setting.
2. Role of the Treating Physician: The treating physician will be responsible for managing participants' medication and medical history but will not be involved in any part of the patient evaluation process, including the assessment of the intervention's effects.

5) Randomization Method

1. Participants meeting the inclusion and exclusion criteria will undergo stratified randomization to ensure balanced distribution.
2. Stratification factors may include gender, age (below 40 years vs. 40 years and older), or disease severity (presence vs. absence of syndesmophytes on X-ray imaging). Final stratification factors will be determined based on the characteristics of enrolled participants.
3. Randomization will be performed by a designated research team member using Microsoft Excel's random function or other randomization software to allocate participants into the Taekwondo training group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with axial spondyloarthritis (axSpA) according to the ASAS classification criteria.
2. Age: Between 19 and 59 years old.
3. Stable medication or non-medication treatment:

   * Patients whose medication regimen has remained stable for at least the past 3 months.
   * Patients who have not taken medication for axSpA for at least the past 3 months.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following conditions:

1. History of orthopedic surgery or fractures within the past 12 months.
2. History of cardiovascular diseases, including ischemic heart disease, cardiomyopathy, heart failure, or stroke.
3. Advanced ankylosis in ankylosing spondylitis, as confirmed by radiographic or CT imaging:

   - Complete ankylosis of at least two regions of the cervical, lumbar, or thoracic spine (i.e., continuous syndesmophyte formation or complete ossification between vertebral bodies).
4. Presence of other musculoskeletal abnormalities or conditions that may limit exercise performance.
5. Diagnosis of cancer within the past 5 years
6. Pregnancy
7. Regular exercise participation within the past 6 months (defined as exercising for at least 60 minutes per session, three or more times per week).
8. Major changes in medication for axial spondyloarthritis during the study period, including:

   1. Initiation or discontinuation of biologic agents or targeted therapies.
   2. Significant changes in the continued use of NSAIDs or sulfasalazine.
   3. Significant changes in the continued use of systemic glucocorticoids.

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score (ASDAS) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) is a composite index that quantifies disease activity in axial spondyloarthritis, incorporating C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR) along with patient-reported outcomes. ASDAS is a continuous measure, with higher scores indicating greater disease activity. Disease activity is classified as follows: ASDAS <1.3 (inactive disease), 1.3-2.1 (low activity), 2.1-3.5 (high activity), and >3.5 (very high activity).
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a self-reported questionnaire designed to assess disease activity in axial spondyloarthritis. It consists of six questions evaluating fatigue, spinal pain, joint pain/swelling, areas of localized tenderness, and morning stiffness (duration and severity).
  Scores range from 0 (no disease activity) to 10 (worst disease activity), with higher scores indicating greater disease activity.
Functional Assessment: Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Bath Ankylosing Spondylitis Functional Index (BASFI) is a self-reported 10-item questionnaire designed to assess functional impairment in patients with axial spondyloarthritis. The questions evaluate activities related to daily living and physical function, including mobility, bending, and the ability to perform tasks. Each item is scored on a 0 to 10 scale, where 0 represents no functional limitation and 10 represents the worst functional limitation.
  Higher BASFI scores indicate greater functional impairment and worse physical function.

SECONDARY OUTCOMES:
Short Form-12 Health Survey Version 2 (SF-12v2) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Short Form-12 Health Survey Version 2 (SF-12v2) is a self-reported measure of health-related quality of life, assessing both physical and mental health across 12 items.
  The survey generates two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), each of which is standardized based on population norms.
  Scores typically range from 0 to 100, with higher scores indicating better health-related quality of life.
Fatigue Severity Scale (FSS) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Fatigue Severity Scale (FSS) is a 9-item self-reported questionnaire that measures the impact of fatigue on daily activities.
  Each item is scored on a 1 to 7 scale, where 1 indicates no fatigue impact and 7 indicates maximum fatigue impact.
  The final score is calculated as the mean of all 9 items, with higher scores indicating greater fatigue severity.
Ankylosing Spondylitis Quality of Life (ASQoL) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire is a self-reported 18-item measure assessing disease-specific quality of life in patients with axial spondyloarthritis.
  Scores range from 0 to 18, with higher scores indicating worse disease-related quality of life.
ASAS Health Index (ASAS-HI) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Ankylosing Spondylitis Assessment Score Health Index (ASAS-HI) is a self-reported questionnaire that assesses overall health status in patients with axial spondyloarthritis.
  The scale consists of 17 dichotomous items (yes/no), with total scores ranging from 0 to 17.
  Higher scores indicate worse health status and greater disease burden.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) is a composite measure of spinal mobility in patients with axial spondyloarthritis.
  It consists of five physical tests evaluating cervical rotation, tragus-to-wall distance, lumbar side flexion, lumbar flexion (modified Schober test), and intermalleolar distance.
  Scores range from 0 (best spinal mobility) to 10 (worst spinal mobility), with higher scores indicating greater spinal stiffness and reduced mobility.
chest expansion | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  Chest expansion will be measured in centimeters (cm) using a standard tape measure.
  The difference between maximal inhalation and maximal exhalation will be recorded at the fourth intercostal space.
  Lower values indicate greater restriction in thoracic mobility.
Numeric Rating Scale (NRS) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Numeric Rating Scale (NRS) is a self-reported measure of pain intensity, where participants rate their pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the worst imaginable pain. Higher scores indicate greater pain intensity.
Body mass index (BMI) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  Body Mass Index (BMI) is calculated as weight in kilograms divided by height in meters squared (kg/m²).
  Higher BMI values indicate greater body mass, with classifications including underweight, normal weight, overweight, and obesity.
waist circumference | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  Waist circumference will be measured in centimeters (cm) using a standard tape measure, with the measurement taken at the midpoint between the lower rib and the iliac crest.
  Higher waist circumference values indicate greater central adiposity, which is associated with increased metabolic risk.
Korean version of the Center for Epidemiologic Studies Depression Scale - Revised (K-CESD-R) | Baseline (Pre-intervention), Week 12 (after RCT), and Week 24 (after control group Taekwondo training)
  The Korean version of the Center for Epidemiologic Studies Depression Scale - Revised (K-CESD-R) is a self-reported 20-item questionnaire designed to assess the severity of depressive symptoms in the general population. Scores range from 0 to 60, with higher scores indicating greater depressive symptom severity.

OTHER OUTCOMES:
Safety Assessments | From enrollment to the end of intervention at 24 weeks
  1. Adverse Events (AEs):
     All unexpected adverse effects related to the intervention will be documented.
  2. Serious Adverse Events (SAEs):
     Any life-threatening events, hospitalizations, or significant health deterioration resulting from the intervention will be recorded.
  3. Non-intervention-related AEs and SAEs:
  All adverse events will be recorded and monitored, even if they are not directly related to the intervention, to ensure the overall safety of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Seoung Wan Nam, M.D., Ph.D., Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data related to primary and secondary outcome measures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after the publication of study results in a peer-reviewed journal. Data will be available for at least 5 years after publication.
Access Criteria: De-identified individual participant data (IPD) related to primary and secondary outcomes, as well as supporting documents (Study Protocol, Statistical Analysis Plan, and ICF), will be available to qualified researchers affiliated with academic or medical institutions. Researchers must submit a formal request, including a study proposal, and access will be granted upon approval by the principal investigator and institution under a data-sharing agreement.
URL: https://wmrc.yonsei.ac.kr/

REFERENCES:
- [Background] Ortolan A, Webers C, Sepriano A, Falzon L, Baraliakos X, Landewe RB, Ramiro S, van der Heijde D, Nikiphorou E. Efficacy and safety of non-pharmacological and non-biological interventions: a systematic literature review informing the 2022 update of the ASAS/EULAR recommendations for the management of axial spondyloarthritis. Ann Rheum Dis. 2023 Jan;82(1):142-152. doi: 10.1136/ard-2022-223297. Epub 2022 Oct 19. PMID 36261247
- [Background] Sveaas SH, Bilberg A, Berg IJ, Provan SA, Rollefstad S, Semb AG, Hagen KB, Johansen MW, Pedersen E, Dagfinrud H. High intensity exercise for 3 months reduces disease activity in axial spondyloarthritis (axSpA): a multicentre randomised trial of 100 patients. Br J Sports Med. 2020 Mar;54(5):292-297. doi: 10.1136/bjsports-2018-099943. Epub 2019 Feb 11. PMID 30745314
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- [Background] O'Dwyer T, O'Shea F, Wilson F. Exercise therapy for spondyloarthritis: a systematic review. Rheumatol Int. 2014 Jul;34(7):887-902. doi: 10.1007/s00296-014-2965-7. Epub 2014 Feb 19. PMID 24549404
- [Background] Wang J, Li X, Yang F, Guo P, Ren C, Duan Z, Zhang Y. Efficacy and safety of mind-body exercise for patients with axial spondyloarthritis: a systematic review and meta-analysis. J Orthop Surg Res. 2024 Sep 28;19(1):586. doi: 10.1186/s13018-024-05072-5. PMID 39342350

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT06823726/Prot_SAP_001.pdf